CLINICAL TRIAL: NCT04730947
Title: Evaluation of the Cardiac and Metabolic Effects of Dapagliflozin in Heart Failure With Preserved Ejection Fraction (CAMEO-DAPA): A Phase II, Prospective, Double-Blind Study
Brief Title: Dapagliflozin (DAPA) Effects in HFpEF
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Barry Borlaug, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20-005646
Record Dates: First submitted 2021-01-27; First posted 2021-01-29 (Actual); Results first posted 2023-10-12 (Actual); Last update posted 2023-10-12 (Actual); Status verified 2023-09

CONDITIONS: Heart Failure With Preserved Ejection Fraction
MeSH Terms: interventions — dapagliflozin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dapagliflozin Group (Experimental): Subjects with HFpEF will take the study drug dapagliflozin daily
  Interventions: Drug: Dapagliflozin
- Placebo Group (Placebo Comparator): Subjects with HFpEF will take a placebo daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dapagliflozin — 10 mg orally once a day
  Arms: Dapagliflozin Group
Drug: Placebo — Taken orally once a day, the placebo looks identical to the study drug but it contains no active ingredient
  Arms: Placebo Group

SUMMARY:
The purpose of this study is to determine whether treatment with Dapagliflozin (DAPA) for 6 months will improve pulmonary capillary wedge pressure (PCWP) during exercise in heart failure/preserved ejection fraction (HFpEF) and improve cardiac metabolism.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent prior to any study specific procedures.
* Male or female.
* Symptoms of dyspnea (NYHA II-III) with no non-cardiac or ischemia explanation.
* EF ≥ 50% + BMI ≥ 30 kg/m^2
* Elevated pulmonary capillary wedge pressure (PCWP) during exercise (≥ 25 mmHg) ascertained at Visit 1. Patients that have consented to study procedures but do not meet this invasive criterion will be considered as screen failures and will not be randomized .

Exclusion Criteria:

* Type I diabetes.
* Type II diabetes with poor control (HgbA1C ≥ 10%).
* Recent hospitalization (< 30 days) or revascularization (< 90 days).
* Primary cardiomyopathy (such as amyloid).
* Constrictive pericarditis.
* Dyspnea due to primary lung disease or myocardial ischemia in the opinion of the investigator.
* Severe anemia (hemoglobin < 9gm/dl.
* Significant left-sided valvular heart disease (> mild stenosis, > moderate regurgitation),
* Severe kidney disease (estimated glomerular filtration rate (GFR) < 30) or liver disease,

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2021-02-24 (Actual); Primary Completion 2022-11-17 (Actual); Study Completion 2022-11-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Barry A Borlaug, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tada A, Burkhoff D, Naser JA, Harada T, Pourmussa B, Reddy YNV, Jensen MD, Carter RE, Demmer RT, Testani JM, Chirinos JA, Borlaug BA. Dapagliflozin Enhances Arterial and Venous Compliance During Exercise in Heart Failure With Preserved Ejection Fraction: Insights From the CAMEO-DAPA Trial. Circulation. 2024 Sep 24;150(13):997-1009. doi: 10.1161/CIRCULATIONAHA.124.068788. Epub 2024 Aug 5. PMID 39101201
- [Derived] Reddy YNV, Carter RE, Sorimachi H, Omar M, Popovic D, Alogna A, Jensen MD, Borlaug BA. Dapagliflozin and Right Ventricular-Pulmonary Vascular Interaction in Heart Failure With Preserved Ejection Fraction: A Secondary Analysis of a Randomized Clinical Trial. JAMA Cardiol. 2024 Sep 1;9(9):843-851. doi: 10.1001/jamacardio.2024.1914. PMID 39046727
- [Derived] Borlaug BA, Reddy YNV, Braun A, Sorimachi H, Omar M, Popovic D, Alogna A, Jensen MD, Carter R. Cardiac and Metabolic Effects of Dapagliflozin in Heart Failure With Preserved Ejection Fraction: The CAMEO-DAPA Trial. Circulation. 2023 Sep 5;148(10):834-844. doi: 10.1161/CIRCULATIONAHA.123.065134. Epub 2023 Aug 3. PMID 37534453
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Groups:
- Dapagliflozin Group: Subjects with heart failure/preserved ejection fraction (HFpEF) will take the study drug dapagliflozin daily
  Dapagliflozin: 10 mg orally once a day
Period: Overall Study
Arm/Group | Dapagliflozin Group | Placebo Group
Started | 21 | 17
Completed | 21 | 16
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dapagliflozin Group | Placebo Group | Total
Number analyzed (Participants) | 21 | 17 | 38
Age, Continuous [Mean (Standard Deviation); unit: years] | 67 (9) | 67 (9) | 67 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 11 | 25
  Male | 7 | 6 | 13
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 21 | 17 | 38

OUTCOME MEASURES:

1. Primary Outcome: Pulmonary Capillary Wedge Pressure (PCWP) at Maximal Exercise
Description: Pulmonary capillary wedge pressure is a measure of cardiac filling pressure, measured using a high-fidelity micromanometer advanced through the lumen of a fluid-filled catheter during exercise.
Time Frame: Baseline, 24 weeks
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Dapagliflozin Group | Placebo Group
Number analyzed (Participants) | 21 | 16
mmHg | -6.6 (7.2) | -0.4 (8.4)
Statistical Analysis 1: Comparison: Dapagliflozin Group vs Placebo Group; Test type: Superiority; p = 0.027, t-test, 2 sided

2. Primary Outcome: Pulmonary Capillary Wedge Pressure (PCWP) at Rest
Description: Pulmonary capillary wedge pressure is a measure of cardiac filling pressure, measured using a high-fidelity micromanometer advanced through the lumen of a fluid-filled catheter during rest.
Time Frame: Baseline, 24 weeks
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Dapagliflozin Group | Placebo Group
Number analyzed (Participants) | 21 | 16
mmHg | -2.5 (3.7) | 1.1 (5.9)
Statistical Analysis 1: Comparison: Dapagliflozin Group vs Placebo Group; Test type: Superiority; p = 0.029, t-test, 2 sided

3. Secondary Outcome: Change in Body Weight
Description: Change in body weight as measured in kilograms (kg)
Time Frame: Baseline, 24 weeks
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Dapagliflozin Group | Placebo Group
Number analyzed (Participants) | 21 | 16
kg | -3.7 (4.2) | -0.2 (2.6)
Statistical Analysis 1: Comparison: Dapagliflozin Group vs Placebo Group; Test type: Superiority; p = 0.006, t-test, 2 sided

4. Secondary Outcome: Change in Total Blood Volume
Description: Total blood volume was assessed using a radiolabeled iodinated albumin (131I, 5-25 μCu) indicator dilution technique with the BVA-100 Blood Volume Analyzer. Measured in millimeters (mL)
Time Frame: Baseline, 24 weeks
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Dapagliflozin Group | Placebo Group
Number analyzed (Participants) | 21 | 16
mL | -118 (542) | 142 (399)
Statistical Analysis 1: Comparison: Dapagliflozin Group vs Placebo Group; Test type: Superiority; p = 0.12, t-test, 2 sided

5. Secondary Outcome: Change in Plasma Volume
Description: Plasma volume was assessed using a radiolabeled iodinated albumin (131I, 5-25 μCu) indicator dilution technique with the BVA-100 Blood Volume Analyzer. Measured in millimeters (mL)
Time Frame: Baseline, 24 weeks
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Dapagliflozin Group | Placebo Group
Number analyzed (Participants) | 21 | 16
mL | -170 (343) | 115 (322)
Statistical Analysis 1: Comparison: Dapagliflozin Group vs Placebo Group; Test type: Superiority; p = 0.014, t-test, 2 sided

6. Secondary Outcome: Change in Right Atrial (RA) Pressure at Maximal Exercise
Description: Right Atrial (RA) pressure is a measure of cardiac filling pressure, measured using a high-fidelity micromanometer advanced through the lumen of a fluid-filled catheter during exercise.
Time Frame: Baseline, 24 weeks
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Dapagliflozin Group | Placebo Group
Number analyzed (Participants) | 21 | 16
mmHg | -3.4 (4.0) | 0.8 (5.6)
Statistical Analysis 1: Comparison: Dapagliflozin Group vs Placebo Group; Test type: Superiority; p = 0.011, t-test, 2 sided

7. Secondary Outcome: Change in Right Atrial (RA) Pressure at Rest
Description: Right Atrial (RA) pressure is a measure of cardiac filling pressure, measured using a high-fidelity micromanometer advanced through the lumen of a fluid-filled catheter during rest.
Time Frame: Baseline, 24 weeks
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Dapagliflozin Group | Placebo Group
Number analyzed (Participants) | 21 | 16
mmHg | -1.6 (2.6) | 0.3 (4.0)
Statistical Analysis 1: Comparison: Dapagliflozin Group vs Placebo Group; Test type: Superiority; p = 0.088, t-test, 2 sided

8. Secondary Outcome: Change in Mean Pulmonary Arterial Pressure (PA) at Maximal Exercise
Description: Pulmonary Arterial (PA) pressure is a measure of cardiac filling pressure, measured using a high-fidelity micromanometer advanced through the lumen of a fluid-filled catheter during exercise.
Time Frame: Baseline, 24 weeks
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Dapagliflozin Group | Placebo Group
Number analyzed (Participants) | 21 | 16
mmHg | -5.2 (6.6) | 0.7 (8.6)
Statistical Analysis 1: Comparison: Dapagliflozin Group vs Placebo Group; Test type: Superiority; p = 0.024, t-test, 2 sided

9. Secondary Outcome: Change in Mean Pulmonary Arterial Pressure (PA) at Rest
Description: Pulmonary Arterial (PA) pressure is a measure of cardiac filling pressure, measured using a high-fidelity micromanometer advanced through the lumen of a fluid-filled catheter during rest.
Time Frame: Baseline, 24 weeks
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Dapagliflozin Group | Placebo Group
Number analyzed (Participants) | 21 | 16
mmHg | -1.8 (4.0) | 1.1 (7.4)
Statistical Analysis 1: Comparison: Dapagliflozin Group vs Placebo Group; Test type: Superiority; p = 0.136, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: Adverse events were collected on each participant from enrollment through approximately one week following the final on-site study visit for a total of approximately seven months.
Arm/Group | Dapagliflozin Group | Placebo Group
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/17
Serious Adverse Events (participants affected / at risk) | 4/21 | 0/17
Other Adverse Events (participants affected / at risk) | 21/21 | 17/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dapagliflozin Group (N=21) | Placebo Group (N=17)
humerus fracture (Surgical and medical procedures) | 1 (1) | 0 (0)
pneumonia related to COVID-19 (Infections and infestations) | 1 (1) | 0 (0)
allergic food reaction (General disorders) | 1 (1) | 0 (0)
hospitalization (General disorders) | 1 (1) | 0 (0) — Hospitalization due to patient not having someone to accompany them to hotel following catheterization
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dapagliflozin Group (N=21) | Placebo Group (N=17)
Minor bruising or bleeding following catheterization (General disorders) | 2 (2) | 2 (2)
Dizziness or dehydration (General disorders) | 8 (8) | 2 (2)
Genitourinary infections (Infections and infestations) | 3 (3) | 1 (1)
Hypoglycemia (General disorders) | 1 (1) | 1 (1)
Worsening dyspenea (General disorders) | 6 (6) | 7 (7)
Worsening fatigue (General disorders) | 3 (3) | 4 (4)
Medication intolerance (General disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-01-13): https://cdn.clinicaltrials.gov/large-docs/47/NCT04730947/Prot_SAP_000.pdf